CLINICAL TRIAL: NCT04825119
Title: Hyperkinetic Movements in Patients With Motor Neuron Disease and in Patients With Spinal Muscular Atrophy and Their Response to Treatment With Nusinersen
Brief Title: Hyperkinetic Movements in Patients With Disease of Motor Neurons and Their Response to Treatment With Nusinersen
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Medical Centre Ljubljana (Other)
Responsible Party: Principal Investigator, Maja Kojović, Principal Investigator, University Medical Centre Ljubljana
Other Study IDs: 0120-293/2019/8/1
Record Dates: First submitted 2021-03-02; First posted 2021-04-01 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Tremor; Involuntary Movements; SMA; MND (Motor Neurone DIsease)
Keywords: Tremor; Minipolymyoclonus; Nusinersen; SMA; MND; ALS
MeSH Terms: conditions — Tremor; Dyskinesias; Amyotrophic Lateral Sclerosis | interventions — nusinersen

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- MND patients: Patients with ''clinically definite ALS'' or ''clinically probable ALS'' or ''clinically probable ALS - laboratory supported'' according to the revised El Escorial diagnostic criteria or with the diagnosis of PMA or PLS will be included.
- SMA patients: SMA patients type I, II, III, and IV will be included.
  Interventions: Drug: Nusinersen

INTERVENTIONS:
Drug: Nusinersen — Patients with SMA who will be treated with nusinersen will be included.
  Other Names: Spinraza
  Groups: SMA patients

SUMMARY:
Hyperkinetic movement disorders in patients with diseases of motor neurons will be studied.

Patients with spinal muscular atrophy (SMA) and motor neuron disease patients will be studied. Involuntary movements will be video recorded and accelerometry with electromyography (EMG) will be recorded in a subset of patients. Hyperkinetic involuntary movements studied will be tremor and minipolymyoclonus. Tremor is defined as involuntary, rhythmic, oscillatory movements of a body part, and minipolymyoclonus are intermittent and irregular movements, with amplitudes sufficient to produce visible movements of the joints. Hyperkinetic movement disorders may be of central or peripheral origin and using accelerometry with EMG may help distinguish the two mechanisms. In patients with SMA the investigators will explore the effect of Nusinersen treatment on phenomenology and amplitude of tremor and minipolymyoclonus.

Aims: To explore the prevalence and phenomenology of hyperkinetic movement disorders in patients with MND and SMA and to study the underlying pathological mechanisms with the use of accelerometry and EMG. To explore the effect of Nusinersen treatment on phenomenology and amplitude of involuntary movements.

Hypotheses: Based on clinical observations the investigators believe it will proven that hyperkinetic movement disorders are common in patients with disease of motor neurons. The investigators hypothesize that hyperkinetic movement disorders in MND and SMA patients are of peripheral origin, being caused by uneven graduation of contraction in the wasted muscles with large motor units being active with no sufficient previous recruitment of small units to smooth contraction of large motor units. If tremor and minipolymyoclonus in SMA are due to the activation of enlarged motor units which are caused by reinnervation of muscle fibers, the treatment with Nusinersen will increase the amplitude of tremor and minipolymyoclonus.

Methods: Presence, quality, and regularity of hyperkinetic movement disorders will be defined using clinical examination, accelerometry and EMG. Hyperkinetic movements will be classified as minipolymyoclonus or tremor. In patients with SMA, the measurements will be repeated 6-12 months after initiation of treatment with Nusinersen.

DETAILED DESCRIPTION:
Background: Minipolymyoclonus and tremor are frequently mentioned as part of the clinical picture of spinal muscular atrophy, but the precise mechanism of the occurrence of tremor and minipolymyoclonus in these patients remains unknown. In the 1970s it was suggested minipolymyoclonus and tremor are caused by reinnervation that follows denervation of muscle fibers in neuropathies. The investigators are not aware of any later or more systematic study on the frequency of minipolymyoclonus and tremor occurrence in SMA patients or its evolution during the disease course. Nusinersen, an antisense oligonucleotide, is a medicine registered for treating SMA. Nusinersen increases the production of the functional survival motor neuron protein by regulating gene expression and thus slows down or stops alpha-motor neuron degradation. MND is considered a disease of upper and lower motor neuron and movement disorders are not considered part of its typical clinical picture. Movement disorders are only reported in MND in association with extrapyramidal or cerebellar degeneration or dysfunction. Contrary to this, the investigators have encountered anecdotal evidence from a number of patients with otherwise typical MND who manifested involuntary jerks and tremor.

Aims: To explore the prevalence and phenomenology of hyperkinetic movement disorders in patients with SMA and MND, to explore the effect of Nusinersen treatment on phenomenology and amplitude of tremor and minipolymyoclonus, and to elucidate the underlying pathological mechanisms by using accelerometry and EMG.

Patients and inclusion/exclusion criteria: All genetically proven SMA patients who will be treated with Nusinersen and consecutive patients followed in MND outpatient clinic will be recruited. Patients with SMA type I, II, III, and IV and patients with ''clinically definite ALS'' or ''clinically probable ALS'' or ''clinically probable ALS - laboratory supported'' according to the revised El Escorial diagnostic criteria or with the diagnosis of PMA or PLS will be included. There will be no exclusion criteria.

Study protocol: All patients will be clinically examined and video-recorded. SMA patients will be examined and video-recorded for the second time 6-12 months after initiation of treatment with Nusinersen. The presence, quality, and regularity of involuntary movements will be evaluated while subjects will be sitting in a chair with hands resting in their lap (usual posture when examining rest tremor), during forward horizontal reach posture, and during finger to nose task. Based on regularity and distribution, hyperkinetic movements will be classified as minipolymyoclonus (MPMC) or tremor. Accelerometry with EMG will be recorded in a subset of patients with hyperkinetic movements.

Methods:

Accelerometry with electromyography: With accelerometry tremor (frequency and amplitude) in the subjects will be objectively evaluated. A triaxle accelerometer will be attached to the 3rd metacarpal bone bilaterally. Simultaneously EMG will be recorded. Bipolar Ag / AgCl surface EMG electrodes will be placed over the flexor carpi radialis and the extensor carpi radialis muscle bilaterally. Electromyography and accelerometry will be recorded while subjects will be sitting in an armchair/wheelchair or lying in a hospital bed (a) at rest position (b) with arms outstretched (postural condition) (c) at the postural condition with 500 g mass attached to the hand (weight loading) and (d) while performing a goal-directed task (action).

Statistical analysis: Clinical measures before and after Nusinersen treatment will be compared using two-related-samples T-test or repeated-measures ANOVA. To assess possible causative mechanisms (disease factors) that determine the presence of involuntary movements, separate multilevel binary logistic analyses will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Genetically proven SMA patients treated with Nusinersen
* ''clinically definite ALS'' or ''clinically probable ALS'' or ''clinically probable ALS - laboratory supported'' according to the revised El Escorial diagnostic criteria or diagnosis of PMA or PLS

Exclusion Criteria:

* No.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Consecutive patients with ALS, PMA, or PLS followed in MND outpatient clinic will be included in the study. Consecutive SMA patients treated with Nusinersen and followed in MND outpatient clinic will be included.
Sampling Method: Probability Sample
Enrollment: 110 (Estimated)
Dates: Start 2017-10-01 (Actual); Primary Completion 2021-07-30 (Estimated); Study Completion 2021-07-30 (Estimated)

PRIMARY OUTCOMES:
Prevalence of involuntary movements in patients with SMA before starting treatment with nusinersen | Baseline (before starting nusinersen treatment)
  All patients will be clinically examined and video-recorded before starting treatment with nusinersen. The presence of involuntary movements will be evaluated as present or not present while subjects will be sitting in a chair with hands resting in their lap (usual posture when examining rest tremor), during forward horizontal reach posture and during finger to nose task.
The effect of nusinersen on the prevalence of involuntary movements in patients with SMA | 6-12 months after starting nusinersen
  All patients will be clinically examined and video-recorded 6-12 months after starting treatment with nusinersen. The presence of involuntary movements will be evaluated as present or not present while subjects will be sitting in a chair with hands resting in their lap (usual posture when examining rest tremor), during forward horizontal reach posture and during finger to nose task.
Characteristics of involuntary movements in patients with SMA before starting treatment with nusinersen | Baseline (before starting nusinersen treatment)
  The quality and regularity of involuntary movements will be evaluated in the standard positons before starting treatment with nusinersen. Based on regularity and distribution, movements observed will be classified as minipolymyoclonus or tremor.
The effect of nusinersen on the characteristics of involuntary movements in patients with SMA | 6-12 months after starting nusinersen
  The quality and regularity of involuntary movements will be evaluated in the standard positons 6-12 moths after starting treatment with nusinersen. Based on regularity and distribution, movements observed will be classified as minipolymyoclonus or tremor.
Amplitude of involuntary movements in patients with SMA before starting treatment with nusinersen | Baseline (before starting nusinersen treatment)
  The quality and regularity of involuntary movements will be evaluated in the standard positons before starting treatment with nusinersen. Accelerometry with EMG will be recorded in all patients with hyperkinetic movements. Amplitude of involuntary movements will be graded on a scale from 0 to 3.
The effect of nusinersen on the amplitude of involuntary movements in patients with SMA | 6-12 months after starting nusinersen
  The quality and regularity of involuntary movements will be evaluated in the standard positons 6-12 moths after starting treatment with nusinersen. Accelerometry with EMG will be recorded in all patients with hyperkinetic movements. Amplitude of involuntary movements will be graded on a scale from 0 to 3.
Prevalence of involuntary movements in patients with MND | Day 1
  Patients will be clinically examined by movement disorders experts and video-recorded. The presence of involuntary movements will be evaluated while subjects will be sitting in a chair with hands resting in their lap (usual posture when examining rest tremor), during forward horizontal reach posture and during finger to nose task.
Characteristics of involuntary movements in patients with MND | Day 1
  The quality and regularity of involuntary movements will be evaluated while subjects will be sitting in a chair with hands resting in their lap (usual posture when examining rest tremor), during forward horizontal reach posture and during finger to nose task. Based on regularity and distribution, hyperkinetic movements will be classified as minipolymyoclonus or tremor.
Amplitude of involuntary movements in patients with MND | Day 1
  In 10 patients accelerometry with electromyography will be recorded at standard positions.

CONTACTS AND LOCATIONS:
Overall Officials: Maja Kojović, PhD, MD, Principal Investigator — University Medical Centre Ljubljana
Locations (1):
- University Medical Centre Ljubljana, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Brooks BR, Miller RG, Swash M, Munsat TL; World Federation of Neurology Research Group on Motor Neuron Diseases. El Escorial revisited: revised criteria for the diagnosis of amyotrophic lateral sclerosis. Amyotroph Lateral Scler Other Motor Neuron Disord. 2000 Dec;1(5):293-9. doi: 10.1080/146608200300079536. No abstract available. PMID 11464847
- [Background] Pupillo E, Bianchi E, Messina P, Chiveri L, Lunetta C, Corbo M, Filosto M, Lorusso L, Marin B, Mandrioli J, Riva N, Sasanelli F, Tremolizzo L, Beghi E; Eurals Consortium. Extrapyramidal and cognitive signs in amyotrophic lateral sclerosis: A population based cross-sectional study. Amyotroph Lateral Scler Frontotemporal Degener. 2015;16(5-6):324-30. doi: 10.3109/21678421.2015.1040028. Epub 2015 May 12. PMID 25967544
- [Background] Dawood AA, Moosa A. Hand and ECG tremor in spinal muscular atrophy. Arch Dis Child. 1983 May;58(5):376-8. doi: 10.1136/adc.58.5.376. PMID 6859919
- [Background] Wurster CD, Ludolph AC. Nusinersen for spinal muscular atrophy. Ther Adv Neurol Disord. 2018 Mar 13;11:1756285618754459. doi: 10.1177/1756285618754459. eCollection 2018. No abstract available. PMID 29568328